CLINICAL TRIAL: NCT05659901
Title: Integrated Prospective and Retrospective Observational Study to Characterize Biomarkers and Disease Progression in Patients With Pelizaeus-Merzbacher Disease
Brief Title: Rocket Study: A Study to Characterize Biomarkers and Disease Progression in Participants With Pelizaeus-Merzbacher Disease
Status: Recruiting | Type: Observational
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NH00005
Record Dates: First submitted 2022-11-22; First posted 2022-12-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pelizaeus-Merzbacher Disease
Keywords: PMD
MeSH Terms: conditions — Pelizaeus-Merzbacher Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pelizaeus-Merzbacher Disease Participants: Participants will undergo CSF collection and neuroimaging procedures, up to Week 106 as a part of prospective study. Each participant's medical and family history data will be collected retrospectively from available medical notes and charts, from birth up to the end of the study period (up to 26 months).

SUMMARY:
The purpose of the study is to prospectively assess longitudinal changes in proteolipid protein 1 (PLP1) protein, disease-related biomarkers in cerebral spinal fluid (CSF) and blood, neuroimaging parameters relevant to Pelizaeus-Merzbacher disease (PMD) and longitudinal changes in performance on clinical, participant, and caregiver-reported outcome assessments to inform the development of therapies for PMD.

DETAILED DESCRIPTION:
This is a multi-center, non-randomized, non-interventional integrated prospective and retrospective study in up to 32 participants with PMD who can undergo general anesthesia or conscious sedation (if necessary) to collect fluid biomarkers (CSF and blood), neuroimaging, and clinical assessments to be used in support of the development of therapies for PMD. The study duration for each participant will be approximately 26 months (Week 106).

ELIGIBILITY:
Inclusion Criteria:

1. Participant has a parent or caregiver capable of providing informed consent (signed and dated) and able to attend all scheduled study visits and provide feedback regarding the participant's symptoms and performance as described in the protocol and be able to comply with all study requirements
2. Participant has a diagnosis of Pelizaeus-Merzbacher Disease with genetic confirmation of PLP1 duplication
3. Male, 6 months-17 years old, inclusive, at the time of informed consent and phenotype consistent with classic PMD
4. No contraindications for lumbar punctures (LPs), blood draws, neuroimaging, sedation (if necessary) or other study procedures

Exclusion Criteria:

1. Clinically significant abnormalities in medical history or physical examination
2. > 2 copies of the PLP1 gene
3. Have any other conditions, which, in the opinion of the investigator would make the participant unsuitable for inclusion, or could interfere with the participant taking part in or completing the study

Ages: 6 Months to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Study Population: Pelizaeus-Merzbacher disease participant population
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Assess Longitudinal Changes in Fluid Biomarkers | Up to 26 months
  Changes in Proteolipid Protein 1 (PLP1) in CSF and disease related biomarkers
Assess Longitudinal Changes in Neuroimaging Parameters | Up to 26 months
  Changes in regional brain volumes (MRI) and in brain metabolites (MRS)
Assess longitudinal changes in performance on clinical, and patient and caregiver-reported outcome assessments | Up to 26 months
  Includes collection of gross and fine motor outcomes, spasticity, dysphagia, cognition and behavior, and sleep.

SECONDARY OUTCOMES:
Characterize health service utilization and economic and disease burden | Up to 26 months

CONTACTS AND LOCATIONS:
Locations (7):
- Ionis Investigative Site, Philadelphia, Pennsylvania, United States
- France (2):
  - Ionis Investigative Site, Clermont-Ferrand
  - Ionis Investigative Site, Le Kremlin-Bicêtre
- Ionis Investigative Site, Göttingen, Germany
- Ionis Investigative Site, Tel Aviv, Israel
- Ionis Investigative Site, Milan, Italy
- Ionis Investigative Site, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.
URL: https://vivli.org/ourmember/ionis/